CLINICAL TRIAL: NCT03113422
Title: Phase II Study of Venetoclax (ABT-199/GDC-0199) in Combination With Obinutuzumab and Bendamustine in Patients With High Tumor Burden Follicular Lymphoma as Front Line Therapy
Brief Title: Phase II Venetoclax, Obinutuzumab and Bendamustine in High Tumor Burden Follicular Lymphoma as Front Line Therapy
Acronym: PrE0403
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE0403; ML39161 (Other: Genentech)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Follicular Lymphoma; Non-Hodgkin's Lymphoma Follicular; Non-Hodgkin's Lymphoma, Adult High Grade
Keywords: High Tumor Burden Follicular Lymphoma; Venetoclax; Obinutuzumab; Bendamustine; Bcl-2 Family Protein Inhibitor; Monoclonal Antibody
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Induction Venetoclax (Experimental): Cycle 1-6: Obinutuzumab intravenously (IV) and bendamustine IV. Cycle 2-6: Venetoclax (oral)
  Interventions: Drug: Induction Venetoclax
- Maintenance Venetoclax (Experimental): Patients with stable or improved disease will receive venetoclax by mouth daily for 24 cycles (1 cycle=1 month) and obinutuzumab IV every 2 months for 12 cycles. Patients with no evidence of disease will receive obinutuzumab IV every 2 months for 12 cycles.
  Interventions: Drug: Maintenance Venetoclax

INTERVENTIONS:
Drug: Induction Venetoclax — 1 cycle = 28 days.
  * Cycle 1-6: Obinutuzumab IV. Cycle 1, Day 1 obinutuzumab 100 mg and Cycle 1, Day 2 obinutuzumab 900 mg for total dose of 1000 mg. On Cycle 1, Day 8 and Day 15 obinutuzumab 1000 mg. Starting with Cycle 2, obinutuzumab 1000 mg on Day 1 only of each cycle.
  * Cycle 1-6: Bendamustine 90 mg/m² IV on Days 1 and 2 of each cycle over 15 minutes after obinutuzumab.
  * Cycle 2-6: Venetoclax 800 mg by mouth daily on Days 1-10 administered before obinutuzumab and/or bendamustine.
  Other Names: GDC-0199; ABT-199; RO5537382
  Arms: Induction Venetoclax
Drug: Maintenance Venetoclax — Patients whose disease is the same or improved will receive venetoclax 800 mg by mouth daily for 24 cycles (1 cycle=1 month) and obinutuzumab 1000 mg IV every 2 months for 12 cycles. Patients with no evidence of disease will receive obinutuzumab 1000 mg IV every 2 months for 12 cycles.
  Other Names: GDC-0199; ABT-199; RO5537382
  Arms: Maintenance Venetoclax

SUMMARY:
Patients with high tumor burden, low grade follicular lymphoma that has never been treated, will receive venetoclax in combination with obinutuzumab and bendamustine.

Venetoclax is an oral Bcl-2 family protein inhibitor. It targets the B-cell lymphoma 2 (BCL-2) protein, which supports cancer cell growth and is overexpressed in many patients with follicular lymphoma. Venetoclax may help to slow down the growth of cancer or may cause cancer cells to die.

The purpose of this study is to see whether adding venetoclax to obinutuzumab and bendamustine improves the response (the tumor shrinks or disappears) in patients with follicular lymphoma.

As of 9/5/2018, a higher than expected incidence of tumor lysis syndrome (TLS) was experienced among patients receiving venetoclax, obinutuzumab and bendamustine on Cycle 1, Day 1 of treatment. TLS is caused by the fast breakdown of cancer cells. These patients developed an increase in some of their blood tests (uric acid, phosphorus, potassium and/or creatinine). They received a medication called rasburicase and continued with treatment. It is unclear if the TLS was due to the venetoclax or the standard treatment of obinutuzumab and bendamustine. For the remaining patients, venetoclax will start on Cycle 2, Day 1 (previously Cycle 1, Day 1).

As of 9/16/2021, additional maintenance therapy has been suspended for those patients who remain on study. These patients will not receive any further treatment and will move on to the two year survival follow-up.

DETAILED DESCRIPTION:
Follicular lymphoma (FL) is the most common low grade lymphoma comprising 70% of low-grade non-Hodgkin's lymphoma (NHL) and 22% of all cases of NHL. The survival rates for patients with indolent NHL remained unchanged from the 1950s through the early 1990s, but recent evidence suggests that outcomes continue to improve. High-risk patients with FL, defined as having advanced stage and high tumor burden have significantly shorter progression free survival despite significant advances.

This is an open-label phase II study of venetoclax in combination with obinutuzumab and bendamustine. Patients will receive induction therapy with obinutuzumab and bendamustine for six cycles (1 cycle = 28 days). Venetoclax will start with 2nd cycle of induction therapy (previously started with cycle 1). There will be a formal, detailed toxicity evaluation after 21 patients complete 3 cycles of treatment.

Patients who achieve partial response or stable disease will receive therapy with obinutuzumab every 2 months for 12 cycles and venetoclax every month for 24 cycles. Patients who achieve a complete response will receive obinutuzumab every 2 months for 12 cycles. Patients with progressive disease will not continue onto the maintenance arm.

Tumor assessments will be performed approximately every 12 weeks during induction and every 6 months during maintenance therapy.

Mandatory pre-treatment tumor tissue sample (i.e., obtained during a previous procedure or biopsy) will be required for research (if sufficient tissue is available). Optional tumor biopsy samples obtained during treatment or post-treatment will also be requested for research.

ELIGIBILITY:
* Patient must have a histologically confirmed (biopsy-proven) diagnosis of follicular B-cell non-Hodgkin lymphoma (WHO classification: follicular center grades 1, 2, and 3a [3b patients are not eligible]), with no evidence of transformation to large cell histology.
* Patient must meet criteria for High Tumor Burden (higher risk) as defined by either the Groupe D'Etude des Lymphomes Follicularies (GELF) criteria [at least one criterion] OR the follicular lymphoma international prognostic index (FLIPI) [score of 3, 4, or 5].
* Patient must have Stage II, III or IV disease.
* Baseline measurements and evaluations (PET/ CT) must be obtained within 10 weeks of randomization to the study. Patient must have at least one objective measurable disease parameter.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Ability to understand and willingness to sign Institutional Review Board (IRB)-approved informed consent.
* Willing to provide mandatory tissue samples (if sufficient tissue available) for research purposes.
* Adequate organ function as measured by the following criteria:

  * Absolute Neutrophil Count (ANC) ≥ 1000/mm³
  * Hemoglobin ≥ 8 g/dL
  * Platelets ˃75,000/mm³
  * Creatinine clearance ≥ 50 mL/min, calculated with the use of 24-hour creatinine clearance or by Cockcroft-Gault formula
  * Total Bilirubin ≤ 1.5x Upper Limit of Normal (ULN) or ≤ 3x ULN for patients with documented Gilbert's syndrome
  * Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 2.5x ULN
  * Alkaline Phosphatase <5x ULN
* All females of childbearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have a blood or urine test to rule out pregnancy within 2 weeks prior to registration.
* Women must not be pregnant or breastfeeding.
* Patient must have had no prior chemotherapy, radiotherapy or immunotherapy for lymphoma. For purposes of this trial, prednisone or other corticosteroids used for non-lymphomatous conditions will not be considered as prior chemotherapy. In addition, a prior/recent short course (<2 weeks) of steroids for symptom relief of lymphoma-related symptoms will not make a patient ineligible.
* Patient must have no recent history of malignancy except for adequately treated basal cell or squamous cell skin cancer, Stage I melanoma of the skin, or in situ cervical cancer. Individuals in documented remission without treatment for ≥ 2 years prior to enrollment may be included at the discretion of the investigator.
* Patient must have no active, uncontrolled infections.
* Patients must be tested for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg+) and hepatitis C (HCV) antibody within 6 weeks of registration. Patients who are chronic carriers of HBV with positive HBsAg+ and positive HCV serology are excluded, as chemotherapy and B-cell depleting therapy have been associated with virus reactivation and fulminant hepatitis. NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) may be included if HBV DNA is undetectable. If enrolled, patients must be willing to undergo monthly HBV DNA testing. Patients with positive HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation.
* HIV positive patients are not excluded, but to enroll, must meet all of the below criteria:

  * HIV is sensitive to antiretroviral therapy.
  * Must be willing to take effective antiretroviral therapy if indicated.
  * No history of CD4 prior to or at the time of lymphoma diagnosis <300 cells/mm³.
  * No history of AIDS-defining conditions.
  * If on antiretroviral therapy, must not be taking zidovudine or stavudine.
  * Must be willing to take prophylaxis for Pneumocystis jiroveci pneumonia during therapy and until at least 2 months following the completion of therapy or until the CD4 cells recover to over 250 cells/mm³, whichever occurs later.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient.
* No major surgery within 2 weeks prior to cycle 1, other than for diagnosis.
* A condition that precludes oral route of administration (venetoclax).
* No known allergies to both xanthine oxidase inhibitors and rasburicase.
* Patient must not require the use of warfarin (because of potential drug-drug interactions that may potentially increase the exposure of warfarin). Blood thinners of other classes are permitted.
* Patient may not receive the following agents within 7 days prior to the first dose of venetoclax:

  * Strong and moderate CYP3A inhibitors
  * Strong and moderate CYP3A inducers
  * Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax.
* Patient must not have serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Portell, MD, Study Chair — University of Virginia
Locations (10):
- United States (10):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of NJ, New Brunswick, New Jersey
  - Fox Chase, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Gunderson Health System Cancer Center, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Result] Portell CA, Jegede OA, Wagner-Johnston N, Nowakowski GS, Fletcher C, Cohen JB, Evens AM, Rosenstein LJ, Craig JW, Reddy N, Kahl BS. Phase II study of venetoclax added to bendamustine and obinutuzumab in patients with high-risk follicular lymphoma as front-line therapy: PrE0403. Blood Cancer J. 2025 May 12;15(1):93. doi: 10.1038/s41408-025-01300-1. PMID 40355425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2017 and November 2020, 56 eligible and treated patients were enrolled.
Pre-assignment Details: Patients were directly assigned to receive induction therapy.
Groups:
- Obinutuzumab + Bendamustine + Venetoclax Induction: Cycle 1-6: Obinutuzumab 1000mg intravenously (IV) Cycle 1-6: Bendamustine 90 mg/m² IV Cycle 2-6: Venetoclax 800 mg by mouth daily on Days 1-10
Period: Overall Study
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients must have histologically confirmed diagnosis of follicular B-cell non-Hodgkin lymphoma; must meet criteria for High Tumor Burden by GELF or FLIPI; Stage II, III, or IV disease; age >=18 years; ECOG PS of 0-2; adequate organ function; must not have had prior chemotherapy, radiotherapy, or immunotherapy for lymphoma; no major surgery within 2 weeks prior to cycle 1.
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 23
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56
Ann-Arbor Stage [Count of Participants; unit: Participants] — Clinically staged, Stage IV is worst stage and indicates extralymphatic organs involvement.
  Participants
    Stage II | 2
    Stage III | 16
    Stage IV | 38
FLIPI-1 Risk Factors [Count of Participants; unit: Participants] — Follicular Lymphoma International Prognostic Index (FLIPI) is a clinical assessment of the number of risk factors present, higher numbers indicates worse prognosis.
  Participants
    0 | 1
    1 | 3
    2 | 20
    3 | 24
    4 | 8
FLIPI-2 Risk Factors [Count of Participants; unit: Participants] — Follicular Lymphoma International Prognostic Index (FLIPI) is a clinical assessment of the number of risk factors present, higher numbers indicates worse prognosis.
  Participants
    0 | 2
    1 | 8
    2 | 19
    3 | 21
    4 | 6
GELF Risk Factors [Count of Participants; unit: Participants] — Groupe d'Etude des Lymphomes Folliculaires (GELF) Criteria/risk factors is a clinical assessment of the number of risk factors present, higher numbers indicates worse prognosis.
  Participants
    0 | 2
    1 | 22
    2 | 15
    3 | 12
    4 | 4
    5 | 1
WHO Disease Stage [Count of Participants; unit: Participants] — WHO disease stage is based on clinical assessment; higher grade indicates worse prognosis.
  Participants
    Grade 1 | 10
    Grade 2 | 32
    Grade 3A | 9
    Missing | 5
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) is a clinical assessment of how disease (cancer) impacts a patient's daily living abilities; higher number indicates greater negative impact on daily living activities.
  Participants
    0 | 35
    1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) at End of Induction
Description: CR assessed in accordance with Lymphoma Response Criteria (Lugano Criteria)
Time Frame: After 6 cycles (at 28 days/cycle) of induction therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
Participants
  Complete Response (CR) | 41
  Partial Response (PR) | 11
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 0
  Unevaluable | 3

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR assessed in accordance with Lymphoma Response Criteria (Lugano Criteria)
Time Frame: After 6 cycles (at 28 days/cycle) of induction therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
Participants
  Yes, Objective Response (CR+PR) | 52
  No, Objective Response (SD+PD+UN) | 4

3. Secondary Outcome: Convert to CR During Maintenance Therapy (From PR in Induction)
Description: Conversion to CR during Maintenance Therapy assessed in accordance with Lymphoma Response Criteria (Lugano Criteria)
Time Frame: Up to 24 cycles which corresponds to 22 months (at 28 days/cycle)
Measure: Count of Participants; unit: Participants
Groups:
- Obinutuzumab + Venetoclax Maintenance: Patients with stable or improved disease will receive venetoclax by mouth daily for 24 cycles (1 cycle=1 month) and obinutuzumab IV every 2 months for 12 cycles. Patients with no evidence of disease will receive obinutuzumab IV every 2 months for 12 cycles.
  Maintenance Venetoclax: Patients whose disease is the same or improved will receive venetoclax 800 mg by mouth daily for 24 cycles (1 cycle=1 month) and obinutuzumab 1000 mg IV every 2 months for 12 cycles. Patients with no evidence of disease will receive obinutuzumab 1000 mg IV every 2 months for 12 cycles.
Arm/Group | Obinutuzumab + Venetoclax Maintenance
Number analyzed (Participants) | 11
Participants
  Complete Response (CR) | 4
  Partial Response (PR) | 3
  Unevaluable | 4

4. Secondary Outcome: Progression-Free Survival (PFS) in the Intent to Treat (ITT) Population.
Description: PFS assessed in accordance with Lymphoma Response Criteria (Lugano Criteria)
Time Frame: Up to 24 months
Measure: Number (90% Confidence Interval); unit: 2-year PFS (% of participants)
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
2-year PFS (% of participants) | 87.5 [75.3 to 93.9]

5. Secondary Outcome: Overall Survival (OS) in the ITT Population.
Description: OS assessed in accordance with Lymphoma Response Criteria (Lugano Criteria)
Time Frame: Up to 24 months
Measure: Number (90% Confidence Interval); unit: 2-year OS (% of participants)
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
2-year OS (% of participants) | 94.6 [86.7 to 97.9]

6. Secondary Outcome: Number of Participants With Treatment-related GRADE 3+ Adverse Events as Assessed by CTCAE V4.0
Description: Number of participants with abnormal laboratory values and/or adverse events related to treatment of GRADE 3 or higher
Time Frame: Adverse events were captured through 6 cycles of therapy (at 28 days/cycle) and for 30 days after the last dose, for a total assessment period of approximately 7 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
Participants | 47

7. Secondary Outcome: Patient Compliance in Receiving Induction Therapy
Description: Off treatment Reasons
Time Frame: Up to 6 cycles (at 28 days/cycle)
Measure: Count of Participants; unit: Participants
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
Number analyzed (Participants) | 56
Participants
  Treatment completed | 34
  Adverse events | 12
  Death | 1
  Investigator discontinued treatment | 5
  Patient withdrawal | 2
  Disease progression | 1
  More than 28 days of treatment interruption | 1

ADVERSE EVENTS:
Time Frame: Adverse events were captured through 6 cycles of therapy (at 28 days/cycle) and for 30 days after the last dose, for a total assessment period of approximately 7 months. Patients were followed for survival for up to 24 months.
Arm/Group | Obinutuzumab + Bendamustine + Venetoclax Induction
All-Cause Mortality (participants affected / at risk) | 3/56
Serious Adverse Events (participants affected / at risk) | 31/56
Other Adverse Events (participants affected / at risk) | 46/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab + Bendamustine + Venetoclax Induction (N=56)
Tumor lysis syndrome (Investigations) | 8 (8)
Back pain (General disorders) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 2 (5)
Nausea (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (4)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vomitting (Gastrointestinal disorders) | 3 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Infusion related reaction (General disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab + Bendamustine + Venetoclax Induction (N=56)
Nausea (Gastrointestinal disorders) | 46 (46)
Fatigue (General disorders) | 34 (34)
Vomitting (Gastrointestinal disorders) | 26 (26)
Diarrhea (Gastrointestinal disorders) | 24 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (23)
Neutropenia (Blood and lymphatic system disorders) | 21 (21)
Headache (General disorders) | 16 (16)
Decreased appetite (Gastrointestinal disorders) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Infusion related reaction (Blood and lymphatic system disorders) | 11 (11)
Hyperuricemia (Renal and urinary disorders) | 10 (10)
AST/ALT increase (Hepatobiliary disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03113422/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03113422/SAP_001.pdf